CLINICAL TRIAL: NCT02291562
Title: Effects of D-9-Tetrahydrocannabinol (THC) and Cannabidiol (CBD) on Human Episodic Memory Function
Brief Title: Effects of THC and CBD on Human Episodic Memory Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LOGIN_EpMem
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tetrahydrocannabinol (Experimental): 10 mg of Tetrahydrocannabinol as capsule (once)
  Interventions: Drug: Tetrahydrocannabinol
- Cannabidiol (Experimental): 600 mg Cannabidiol capsule (once)
  Interventions: Drug: Cannabidiol
- placebo (Placebo Comparator): placebo capsule (once)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Tetrahydrocannabinol — 10 mg Tetrahydrocannabinol (capsule, once) oral intake
  Arms: Tetrahydrocannabinol
Drug: Cannabidiol — 600 mg Cannabidiol (capsule, once) oral intake
  Arms: Cannabidiol
Drug: placebo — placebo (capsule, once) oral intake
  Arms: placebo

SUMMARY:
THC and CBD have distinct symptomatic and behavioral effects. In healthy individuals, THC can induce psychotic symptoms and anxiety, and can impair memory. In contrast, CBD has anxiolytic and possibly antipsychotic properties, while not impairing memory and other cognitive functions. Instead, CBD has been shown to have significant neuroprotective effects. In humans, CBD values correlated positively with gray matter concentration in bilateral hippocampus. Recent data from experimental animals and in vitro studies suggest that these distinct effects might be caused by opposing effects on brain cannabinoid receptors.

Neuroimaging studies have consistently identified brain activity recorded at prefrontal and medial temporal regions as relevant for episodic memory. Additionally, the abundance of cannabinoid receptors in the hippocampus and the parahippocampal and entorhinal cortices suggests a potential impact of CBD in memory deficits typical in healthy aging. However, the evidence relating cannabinoids to these conditions is relatively recent and has been obtained from either biochemical or pharmacological studies. It might be hypothesized that CBDs could be useful to delay or even arrest the progression of functional and structural neuronal degeneration.

The investigators will use an episodic memory paradigm to test the effects of THC, CBD and placebo on memory encoding and retention and the underlying neuronal networks on healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* no acute or chronic disease

Exclusion Criteria:

* opioid intake
* medication or drug abuse
* kidney or liver dysfunction
* claustrophobia
* none removable metallic parts (e.g. hip replacement)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in BOLD (blood oxygen level dependent) responses | immediate
  Differential changes of the BOLD response under the three different conditions (THC, CBD, placebo) during the learning and the test phase of the memory paradigm

SECONDARY OUTCOMES:
Changes in behavioral measures | immediate
  Differential changes in reaction times and number of correct responses during the three different conditions (THC, CBD, placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Grimm, M.D., Study Chair — Central Institute of Mental Health
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany